CLINICAL TRIAL: NCT06153849
Title: Analyzing the Urine Microbiome and Chromosomal Instability by Whole Genome Sequening in Bladder Cancer Patients During BCG Instillation for Disease Follow-up
Brief Title: Analyzing the Urine During BCG Instillation in Bladder Cancer Patients for Disease Followup
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Shuxiong Zeng, M.D., Ph.D, Changhai Hospital
Other Study IDs: CH-LC-WGS-BCGinstillation
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Urine biomarker; Microbiome; Bacillus Calmette-Guérin instillation; Chromosomal instability; Low coverage whole genome sequencing
MeSH Terms: conditions — Urinary Bladder Neoplasms; Chromosomal Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples were collected form bladder cancer patient and DNA was extracted from urine sediment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BCG instillation patient: Patients with pathology-confirmed median to high risk urothelial carcinoma defined by 2023 EAU guideline, underwent transurethral resection of bladder tumor and receiving BCG instillation therapy.
  Interventions: Diagnostic Test: urine sample collection

INTERVENTIONS:
Diagnostic Test: urine sample collection — Urine samples from patients receiving BCG instillation was collected for LC-WGS to evaluate CIN and urinary microbiome.

SUMMARY:
Bacillus Calmette-Guerin (BCG) has been extensively utilized in intravesical instillation therapy for patients with medium to high risk non-muscle invasive bladder cancer (NMIBC) following transurethral resection of bladder tumor (TURBT). Nevertheless, the efficacy of BCG instillation can fluctuate between patients, with 40.5% experiencing disease recurrence during BCG therapy. The effectiveness of BCG instillation may be linked to the urinary microbiome and immune microenvironment. Additionally, small residual lesions post-TURBT could also result in bladder cancer recurrence. Low coverage whole genome sequencing (LC-WGS) can be used to detect the urinary microbiome and chromosomal instability (CIN), making it feasible to predict the recurrence or progression of bladder cancer during BCG instillation therapy. Here, we intend to evaluate the feasibility of detecting urine samples of bladder cancer patients receiving BCG instillation to predict the bladder cancer recurrence.

DETAILED DESCRIPTION:
NMIBC at medium to high risk showcases a recurrence rate of 40.5% post-TURBT, thus necessitating frequent monitoring and bladder instillation. Among patients with medium to high-risk NMIBC, the preferred treatment is BCG. The high recurrence rate of this illness is associated with BCG's effectiveness and residual cancer, yet the full understanding of BCG installation's mechanism complicates the prediction of its efficacy among individuals with bladder cancer.

Previously, it was believed that the urinary system was sterile; however, recent high-throughput sequencing and enhanced quantitative urine culture have confirmed the presence of resident bacteria in the urine of healthy individuals. Microorganisms within the bladder have the potential to alter the immune microenvironment, consequently impacting the efficacy of BCG instillation.

CIN denotes continuous errors in chromosome separation during cell division, encompassing numerical and structural instability. Loss of the Y chromosome (LOY) represents a specific type of CIN associated with cancer prognosis. CIN serves as a hallmark of malignancies and can be employed to indicate the presence of minimal residual disease (MRD) subsequent to TURBT. Analyzing LOY can better elucidate the disease's progression, and more exploration is necessary to comprehend the significance of detecting CIN for predicting tumor recurrence.

LC-WGS is a cost-effective, efficient, and robust technique that can be used to analyze both microorganism and human genomes in urine samples. The microbiome is commonly detected using 16S ribosomal sequencing. Compared to 16S sequencing, LC-WGS provides advantages such as enhanced detection of bacterial species, diversity, and improved gene prediction. In the context of CIN and LOY detection, LC-WGS technology offers heightened sensitivity, low cost, and high throughput compared to traditional methods such as comparative genomic hybridization or fluorescence in situ hybridization.

In this prospective, single-arm observational clinical trial, the investigators aim to evaluate LOY, CIN, and the urinary microbiome detected by LC-WGS for the assessment of BCG instillation efficacy and NMIBC follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 18 years and signed informed consent form.
* Participants diagnosed with median to high risk NMIBC underwent TURBT and received BCG instillation therapy.

Exclusion Criteria:

* Participants with urinary tract infection
* Antibiotic treatment within the last month
* Immuno- /chemo- therapy within the past 6 months
* Immunosuppressive therapy
* Indwelling urinary catheter
* Additional major diagnosis known to affect the gut or bladder microbiota (e. g. liver cirrhosis, systemic sclerosis, inflammatory bowel disease, inflammatory bowel syndrome, celiac disease, neuropathic bladder)
* Participants with urothelial carcinoma accompanied by other malignancy.
* Individuals unwilling to sign the consent form or unwilling to provide urine sample for test or quality of urine sample is poor.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with medianl to high risk NMIBC underwent TURBT and received BCG instillation therapy in Changhai Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between urinary microbiome and BCG instillation efficacy. | through study completion, an average of 1 year
  Comparison of urinary microbiome between relapsed and non-relapsed patients during follow-up.

SECONDARY OUTCOMES:
Correlation between LOY and prognosis. | through study completion, an average of 1 year
  Comparison of LOY event frequency between relapse patients and non-relapse patients during follow-up.
Correlation between CIN and tumor relapse | through study completion, an average of 1 year
  Comparison of MRD reflected by CIN level in urine samples between relapsed and non-relapsed patients during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not public for privacy protection purpose. Data without private information may be provided on request.

REFERENCES:
- [Background] Sansregret L, Vanhaesebroeck B, Swanton C. Determinants and clinical implications of chromosomal instability in cancer. Nat Rev Clin Oncol. 2018 Mar;15(3):139-150. doi: 10.1038/nrclinonc.2017.198. Epub 2018 Jan 3. PMID 29297505
- [Background] Krajewski W, Zdrojowy R, Grzegolka J, Krajewski P, Wrobel M, Luczak M, Kolodziej A. Does Mantoux Test Result Predicts BCG Immunotherapy Efficiency and Severe Toxicity in Non-Muscle Invasive Bladder Cancer. Urol J. 2019 Oct 21;16(5):458-462. doi: 10.22037/uj.v0i0.4542. PMID 30471076
- [Background] Babjuk M, Burger M, Capoun O, Cohen D, Comperat EM, Dominguez Escrig JL, Gontero P, Liedberg F, Masson-Lecomte A, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Seisen T, Soukup V, Sylvester RJ. European Association of Urology Guidelines on Non-muscle-invasive Bladder Cancer (Ta, T1, and Carcinoma in Situ). Eur Urol. 2022 Jan;81(1):75-94. doi: 10.1016/j.eururo.2021.08.010. Epub 2021 Sep 10. PMID 34511303
- [Result] Ranjan R, Rani A, Metwally A, McGee HS, Perkins DL. Analysis of the microbiome: Advantages of whole genome shotgun versus 16S amplicon sequencing. Biochem Biophys Res Commun. 2016 Jan 22;469(4):967-77. doi: 10.1016/j.bbrc.2015.12.083. Epub 2015 Dec 22. PMID 26718401
- [Result] Han RF, Pan JG. Can intravesical bacillus Calmette-Guerin reduce recurrence in patients with superficial bladder cancer? A meta-analysis of randomized trials. Urology. 2006 Jun;67(6):1216-23. doi: 10.1016/j.urology.2005.12.014. PMID 16765182